CLINICAL TRIAL: NCT02177331
Title: Lacidipine in Medical Practice: Incidence of Rare Adverse Drug Reactions During Long-term Treatment. 3rd Follow-up Study - Long-term Use in the 4th and 5th Year Treatment Years
Brief Title: Lacidipine in Medical Practice in Patients With Mild to Moderate Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 231.215
Record Dates: First submitted 2014-06-24; First posted 2014-06-27 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — lacidipine

ARMS (1):
- Lacidipine (Experimental)
  Interventions: Drug: Lacidipine

INTERVENTIONS:
Drug: Lacidipine

SUMMARY:
In order to confirm the proposed metabolic effect of lacidipine these follow-up study was to provide long-term data on its impact on liver function, glucose homoeostasis and lipid metabolism. Additionally, its adverse drug reactions and antihypertensive effects were to be studied.

ELIGIBILITY:
Inclusion Criteria:

* Fulfillment of entry criteria for the preceding yearly study
* Male or female patients aged between 20 and 85 years
* Known history of mild to moderate essential hypertension requiring drug treatment, WHO grade I to II
* Controlled blood pressure (RR diastolic ≤ 90 mm Hg or 91 - 95 mm Hg and concurrent reduction in blood pressure of at least 10 mm compared to baseline level) during treatment with lacidipine at a dose of 2 - 6 mg once a day
* Final visit of the previous yearly study (Visit 4) completed as scheduled
* Informed consent to participate in the follow-up study

Exclusion Criteria:

* Violation of entry/exclusion criteria on enrolment in the preceding yearly study
* Occurrence of the following exclusion criteria in the intervening period:

  * Pregnancy, lactation, possibility of conception without the use of a scientifically recognised method of contraception
  * Secondary form of hypertension
  * Consumptive illness
  * Clinically manifest concomitant cardiovascular illness, e.g.: aortic or mitral valve stenosis, hypertrophic obstructive cardiomyopathy or any other condition hindering left ventricular outflow, aortic isthmus stenosis, severe (NYHA Class III or higher) or decompensated heart failure, clinically relevant hypo- or hyperkinetic cardiac arrhythmia
  * Myocardial infarction or cerebrovascular accident within the 6 months prior to the start of the follow-up study
  * Hypersensitivity to dihydropyridines
  * Concomitant long-term treatment (> 3 weeks) with antihypertensive substances not envisaged in the protocol (exception: short-acting nitrates), sedatives, tricyclic antidepressants
  * Suspected alcohol, narcotic or drug abuse

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 1995-06; Primary Completion 1998-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with rare adverse drug reactions | up to 24 months
Change in alkaline phosphatase (AP) | up to 24 months
Change in serum glutamic - pyruvic transaminase (SGPT) | up to 24 months

SECONDARY OUTCOMES:
Change in serum glutamic - oxaloacetic transaminase (SGOT) | up to 24 months
Number of patients with abnormal changes in laboratory parameters | up to 24 months
Changes in systolic and diastolic blood pressure | up to 24 months
Changes in gamma glutamyl transferase (gamma-GT) | up to 24 month